CLINICAL TRIAL: NCT06453512
Title: A Study to Evaluate the Emollient Performance of Doublebase Once in the Treatment of Atopic Eczema Using SCORAD, Patient Questionnaires and Skin Hydration Measurements
Brief Title: A Study to Evaluate the Emollient Performance of Doublebase Once in the Treatment of Atopic Eczema
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dermal Laboratories Ltd (Industry)
Collaborators: Nottingham University Hospitals NHS Trust (Other); Sherwood Forest Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DLPF-01
Record Dates: First submitted 2024-05-31; First posted 2024-06-11 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Atopic Eczema
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Post market Surveillance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Main Study (Other): Main Study which also involves the subgroup
  Interventions: Device: Doublebase Once

INTERVENTIONS:
Device: Doublebase Once — Emollient

SUMMARY:
A 4 week, open label, multi-centre (GP setting), post market clinical follow-up study with Doublebase Once in patients of any age and any severity of atopic eczema.

The study will involve patients who are already using emollients as part of their treatment regime, switching to Doublebase Once. Patients will ideally apply the product once daily for 4 weeks and SCORAD assessments will be performed, and patient questionnaires will be completed. A subgroup of adult patients (up to 15 patients) will also undergo skin hydration measurements for the first 8 days to evaluate objective measurements of skin hydration in patients with atopic eczema.

Photographs of the same, representative area of eczema will also be taken for all patients at baseline and after 4 weeks of using Doublebase Once.

DETAILED DESCRIPTION:
This is a prospective, open label, uncontrolled study which will be performed in multiple GP centres, in patients of all ages, who have any severity of atopic eczema. It is anticipated that approximately 75 patients will need to be screened to enrol 65 eligible patients and to complete the study with 50 evaluable patients. This study is being conducted as part of the manufacturer's undertaking to follow up the clinical performance of the device in the post marketing phase (Post Marketing Clinical Follow-up (PMCF)). It will provide additional quantitative information on the product in a real-world environment in various age groups and severities of atopic eczema using validated assessment methods and patient feedback.

Study patients will be asked to use Doublebase Once only once daily for 4 weeks, instead of their usual emollient. If they need to use Doublebase Once more frequently, this will be recorded in their patient diaries, as will any other topical or systemic treatments that they may need to use during the study period (e.g. corticosteroids). Patients will also be able to use Doublebase Once as a soap substitute.

A SCORAD assessment will be performed by the investigator/ research nurse at baseline and then after 1 and 4 weeks of treatment. Patients or their parents/ legal guardians will be asked to complete questionnaires at baseline and after 4 weeks of treatment.

A subgroup of adult patients (of up to 15 patients) will have additional skin hydration measurements (corneometry) taken before switching emollient to Doublebase Once and on 4 more occasions during the first 8 days to evaluate changes in skin hydration in patients with atopic eczema, this will be performed at the same, representative, predetermined selected area of eczema. Measurements will be taken in triplicate (and the mean calculated) and each reading and the mean value will be documented in the patients CRF at baseline, 24 hours after the first application and then again on days 3, 5 and 8 (prior to the application for that day). This subgroup will then continue in the study for the SCORAD and questionnaire follow-up at the same visit timings as the rest of the study population (see 7.12.1.1).

Photographs of one eczema affected area, which will not include any recognisable or identifiable features, private areas or details of the patient, will also be taken at baseline and again after 4 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* ii) Patients with atopic eczema (personal history or combined personal and familial atopy), of any severity in accordance with the NICE categorisation set out in the table below.

iii) Baseline SCORAD assessment score of at least 15. iv) Patients or their parents/ legal guardians must be able to read and understand the patient information sheet and sign the Consent Form/Assent Form.

v) Patients normally managing their eczema by regular and ongoing use of leave-on emollient(s).

vi) Patients who are not currently using systemic or topically applied antibiotics or Doublebase Once.

vii) Patients who are willing to use Doublebase Once, once daily, as their only leave-on emollient, for 4 weeks.

viii) Patients who are willing to continue to use their standard cleansing regime and/or Doublebase Once as a soap substitute for the duration of the study.

Additional inclusion criterion for subgroup for skin hydration assessments:

i) Baseline corneometry measurement of ≤40 arbitrary units.

Exclusion Criteria:

i) Are currently using or have used in the previous month, any systemic or topically applied antibiotics or Doublebase Once for their atopic eczema.

ii) Have a known history of intolerance or skin sensitivity to any of the ingredients of Doublebase Once (as identified on the patient information sheet and product labelling), or similar products.

iii) Currently participating in any other ongoing research studies or have participated in a study in the previous 30 days.

iv) Patients, or their parents/ legal guardians, who may have difficulties completing the questionnaire, which will be written in English only.

v) Employees of the Sponsor or Investigators, or any immediate family member (partner, offspring, parents, siblings, or sibling's offspring) of such employees.

vi) Patients with any medical condition which, in the opinion of the Investigator, may adversely influence their ability to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in SCORAD after 4 weeks of treatment | 4 weeks
  The SCORAD scoring is described in section 7.4.1. For each patient, a score will be obtained at baseline, after 4 weeks. The minimum score is 0 (best outcome) and the maximum score is 103 (worst outcome). The change score will be calculated by subtracting the baseline score from the score after 4 weeks. The actual scores after 4 weeks and the change from baseline will be summarised using summary statistics. In addition, the change from baseline will be presented with a 95% confidence interval (CI), and the following hypotheses will be tested at the two-sided 5% significance level using a paired t-test.
  The SCORAD score is from 0-103 and there is a minimum score of 15 at inclusion. A reduction in total score represents an improvement in the overall condition.

SECONDARY OUTCOMES:
Change from baseline in SCORAD after 1 week of treatment. | 1 week
  The change from baseline in SCORAD after 1 week of treatment will be summarised and analysed in the same way as the primary endpoint.
  The SCORAD score is from 0-103 and there is a minimum score of 15 at inclusion. A reduction in total score represents an improvement in the overall condition.
SCORAD individual items | 4 weeks
  Individual items of the SCORAD will be summarised using descriptive statistics (frequencies for categorical items and summary statistics for continuous measures). These items will be formally evaluated using inferential statistics by comparing values after weeks 1 and 4 versus baseline. The redness, dryness and swelling scores at week 4 will be compared to baseline using an ordinal logistic regression model for paired data. The odds of being in a better outcome category post-treatment compared to pre-treatment will be calculated with a 95% CI and p-value. The itch and sleeplessness scores post-treatment will be compared to the pre-treatment value using a paired t-test, or a Wilcoxon signed rank test if assumptions of Normality are violated. Change from baseline itch and sleeplessness (separately) will be presented with a 95% CI.
Patient Questionnaire | 4 weeks
  For each of the five quality of life questions and for the sum score from the five questions, the score post-treatment will be compared to the pre-treatment value using a paired t-test.
  The Patient Questionnaire (QoL) score is calculated at baseline and a reduction in total score overall represents a Patient perceived improvement in the overall condition.
Skin Hydration | 8 days
  Skin hydration assessments will be performed in up to 15 adults and are a subgroup of the main study. The corneometry values at each visit and the change from baseline will be summarised using summary statistics. The area under the curve (AUC) over the assessment period up to Day 8 will be calculated using the trapezoidal rule.

OTHER OUTCOMES:
Correlation between SCORAD and corneometry | 8 days
  The correlation between change from baseline in SCORAD and change from baseline in corneometry will be assessed in the skin hydration subgroup using the values recorded on Day 8. The Spearmank rank correlation will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Simon T Royal, BMedSci BM BS, Principal Investigator — Dermal Laboratories Ltd
Locations (1):
- Cripps Medical Centre, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No